CLINICAL TRIAL: NCT05272774
Title: Efficacy of the FOREST+ Stress Recovery Program for Healthcare Workers: A Randomized Controlled Trial
Brief Title: Stress Recovery Program FOREST+ for Healthcare Workers
Acronym: FOREST+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25 / (1.3) 250000-KP-22-II
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-02

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Forests

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated either to the intervention or control groups. The control group will use the intervention without feedback from therapist but with support on-demand. The control group will participate in the program at the same time as the intervention group with therapist support.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a 6-week online stress recovery intervention with the support from therapist.
  Interventions: Behavioral: FOREST+
- Control group (Experimental): The control group will use the intervention with on-demand support. The control group will participate in the program at the same time as the intervention group.
  Interventions: Behavioral: FOREST+

INTERVENTIONS:
Behavioral: FOREST+ — The intervention will be delivered as an online stress recovery intervention consisting of six weekly modules. Modules include an introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. These modules have been chosen after considering the themes that could be most useful for healthcare workers under high stress. Each module consists of a psychoeducational and an exercise component.

SUMMARY:
The aim of the study is to assess the efficacy of an online stress recovery intervention for healthcare workers receiving therapist-assisted or on-demand support.

DETAILED DESCRIPTION:
The intervention will be delivered as an online stress recovery program for healthcare workers, consisting of six modules. Modules include an introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. These modules have been chosen after considering themes that could be most useful for healthcare workers under high stress. Each module consists of a psychoeducational and an exercise component. During the program, a therapist provides individual feedback on the exercises completed and can also be available on request.

The effect of the intervention will be compared with a control group that will use the program with support on-demand. The intervention will be delivered in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* licensed healthcare professionals currently working under license;
* at least 18 years old;
* comprehending Lithuanian language;
* access to internet.

Exclusion Criteria:

* acute psychiatric crisis;
* high suicide risk;
* interpersonal violence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Change on Recovery Experience Questionnaire | Pre-treatment, post-treatment, 3 months follow-up
  Changes on stress recovery are measured. Recovery Experiences Questionnaire (Sonnentag & Fritz, 2007) is a self-report measure consisting of 16 questions. All items are answered on a 5-point Likert scale ranging from 1 (Totally disagree) to 5 (Totally agree). A higher score indicates more pronounced recovery.

SECONDARY OUTCOMES:
Change on Perceived Stress Scale | Pre-treatment, post-treatment, 3 months follow-up
  Changes on perceived stress are measured. Perceived Stress Scale (PSS-10, Cohen et al., 1983) is a self-report measure and consists of 10 questions. All items are answered on a 5-point Likert scale that ranges from 0 (Never) to 4 (Very often). Higher score indicates more pronounced perceived stress.
Change on Patient Health Questionnaire | Pre-treatment, post-treatment, 3 months follow-up
  Changes on depression symptoms are measured. Patient Health Questionnaire-9 (PHQ-9, Kroenke et al., 2001) is a self-report measure and consists of 9 questions. All items are answered on a 4-point Likert scale that ranges from 0 (Not at all) to 3 (Nearly every day). Higher score indicates more pronounced depression symptoms.
Change on Generalized Anxiety Disorder Questionnaire | Pre-treatment, post-treatment, 3 months follow-up
  Changes on anxiety symptoms are measured. Generalized Anxiety Disorder Questionnaire-7 (GAD-7, Kroenke et al., 2001) is a self-report measure and consists of 7 questions. All items are answered on a 4-point Likert scale that ranges from 0 (Not at all) to 3 (Nearly every day). Higher score indicates more pronounced anxiety symptoms.
Change on Well-being Index | Pre-treatment, post-treatment, 3 months follow-up
  Changes on well-being are measured. Well-being Index (WHO-5, Bech, 2004) is a self-report measure and consists of 5 questions. All items are answered on a 6-point Likert scale that ranges from 0 (At no time) to 5 (All of the time). Higher score indicates more pronounced well-being.
Change on Moral Injury Outcome Scale | Pre-treatment, post-treatment, 3 months follow-up
  Changes on moral injury are measured. Moral Injury Outcome Scale (MIOS, Litz et al., 2020) is a self-report measure and consists of 15 questions. All items are answered on a 5-point Likert scale that ranges from 0 (Strongly disagree) to 4 (Strongly agree). Higher score indicates more pronounced moral injury.

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Kazlauskas, Ph.D., Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No